CLINICAL TRIAL: NCT01631474
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Vehicle-Controlled, Dose Escalating Study to Evaluate the Safety and Efficacy of Cortexolone 17a-Propionate (CB-03-01) Cream Applied Once or Twice-Daily for 12 Weeks in Subjects With Facial Acne Vulgaris
Brief Title: A Phase 2 Dose Escalating Study to Evaluate the Safety and Efficacy of CB-03-01 Cream in Subjects With Facial Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intrepid Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 171-7151-201
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Results first posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-10

CONDITIONS: Acne Vulgaris
Keywords: acne; anti-androgen; clascoterone; cassiopea
MeSH Terms: conditions — Acne Vulgaris | interventions — Clascoterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Low-dose active, BID (Experimental): low dose of CB-03-01, 0.1% applied twice a day
  Interventions: Drug: CB-03-01
- Medium-dose active, BID (Experimental): medium dose of CB-03-01, 0.5% applied twice a day
  Interventions: Drug: CB-03-01
- High-dose active, QD (Experimental): high dose of CB-03-01, 1% applied once a day
  Interventions: Drug: CB-03-01
- High-dose active, BID (Experimental): high dose of CB-03-01, 1% applied twice a day
  Interventions: Drug: CB-03-01
- Vehicle, QD or BID (Placebo Comparator): vehicle cream, applied once or twice a day
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: CB-03-01 — Topical cream, applied once a day
  Other Names: clascoterone
  Arms: High-dose active, QD
Drug: Vehicle — Topical cream, applied once or twice a day
  Arms: Vehicle, QD or BID
Drug: CB-03-01 — Topical cream, applied twice a day
  Other Names: clascoterone
  Arms: High-dose active, BID; Low-dose active, BID; Medium-dose active, BID

SUMMARY:
CB-03-01 is being developed for the topical treatment of acne vulgaris, an androgen-dependent skin disorder. The purpose of this study is to compare the safety and efficacy of multiple concentrations of CB-03-01 to vehicle in the treatment of acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or non-pregnant female. Females must be post-menopausal, surgically sterile or using highly effective birth control methods.
* Subject has provided written and verbal informed consent/assent.
* Subject has facial acne vulgaris (including the nose).
* Subject is willing to comply with study instructions and return to the clinic for required visits.
* Subject has used the same type and brand of make-up, other facial products (including cleanser) and hair products (e.g., shampoo, gel, hair spray, mousse, etc.) for at least one month prior to the study start and agrees to continue his/her other general skin and hair care products and regimen for the entire study.

Exclusion Criteria:

* Subject is pregnant, lactating, or is planning to become pregnant during the study.
* Subject is currently enrolled in an investigational drug or device study.
* Subject has received an investigational drug or been treated with an investigational device within 30 days prior to the study start.
* Subject has the need or plans to be exposed to artificial tanning devices or excessive sunlight during the trial
* Subject has used any of the following topical anti-acne preparations or procedures on the face:

  * Topical anti-acne treatments including but not limited to over-the-counter acne cleaners or treatments, benzoyl peroxide, antibiotics, azelaic acid, sulfa based products, corticosteroids and salicylic acid within two weeks of the initiation of treatment.
  * Retinoids, including tazarotene, adapalene, tretinoin, within four weeks of the initiation of treatment.
  * Light treatments, microdermabrasion or chemical peels within eight weeks of the initiation of treatment.
* Subject has used the following systemic anti-acne medications:

  * Corticosteroids (including intramuscular and intralesional injections) within four weeks of the initiation of treatment. Inhaled, intranasal or ocular corticosteroids are allowed if use is stable (stable use is defined as dose and frequency unchanged for at least four weeks prior to the initiation of treatment).
  * Antibiotics within four weeks of the initiation of treatment with the exception of five days or less of antibiotic therapy during this period, but with no antibiotics use permitted within one week prior to the initiation of treatment.
  * Spironolactone within eight weeks of the initiation of treatment with the exception of five days or less of spironolactone therapy during this period, but with no spironolactone use permitted within one week prior to the initiation of treatment.
  * Retinoid therapy within six months of the initiation of treatment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R&D Cassiopea, Study Director — Cassiopea S.p.A.
Locations (13):
- United States (13):
  - Dermatology Research Associates, Los Angeles, California
  - Therapeutics Clinical Research, San Diego, California
  - University Clinical Trials, San Diego, California
  - International Clinical Research - US, LLC, Sanford, Florida
  - Gwinnett Clinical Research Center, Inc., Snellville, Georgia
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Indiana Clinical Trials Center, Plainfield, Indiana
  - Marina I. Peredo, M.D., PC, Smithtown, New York
  - Penn State Milton S. Hershey Medical Center - Dept. of Dermatology, Hershey, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - J & S Studies, College Station, Texas
  - UT Houston Health Science Center, Houston, Texas
  - Virginia Clinical Research, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low-dose Active, BID | Medium-dose Active, BID | High-dose Active, QD | High-dose Active, BID | Vehicle, QD or BID
Started | 72 | 76 | 70 | 70 | 75
Completed | 58 | 64 | 61 | 59 | 62
Not Completed | 14 | 12 | 9 | 11 | 13
Not completed — Lost to Follow-up | 8 | 5 | 7 | 5 | 5
Not completed — Withdrawal by Subject | 4 | 4 | 2 | 6 | 5
Not completed — Lack of Efficacy | 2 | 2 | 0 | 0 | 2
Not completed — Noncompliance with Study Drug | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population. The ITT population included all subjects enrolled in the study who were randomized and dispensed test article.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-dose Active, BID | Medium-dose Active, BID | High-dose Active, QD | High-dose Active, BID | Vehicle, QD or BID | Total
Number analyzed (Participants) | 72 | 76 | 70 | 70 | 75 | 363
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.8 (5.77) | 20.4 (6.31) | 18.3 (6.14) | 21.0 (6.22) | 19.2 (5.25) | 19.7 (5.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 42 | 38 | 37 | 43 | 196
  Male | 36 | 34 | 32 | 33 | 32 | 167
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 20 | 6 | 15 | 13 | 76
  Not Hispanic or Latino | 50 | 56 | 64 | 55 | 62 | 287
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 2 | 0 | 3
  Asian | 1 | 3 | 4 | 4 | 4 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1 | 2
  Black or African American | 12 | 14 | 16 | 20 | 12 | 74
  White | 58 | 54 | 50 | 42 | 53 | 257
  More than one race | 1 | 2 | 0 | 2 | 4 | 9
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 2
Baseline IGA [Count of Participants; unit: Participants]
  0 - Clear | 0 | 0 | 0 | 0 | 0 | 0
  1 - Almost clear | 0 | 0 | 0 | 0 | 0 | 0
  2 - Mild | 10 | 6 | 15 | 18 | 11 | 60
  3 - Moderate | 56 | 62 | 44 | 32 | 53 | 247
  4 - Severe | 6 | 8 | 11 | 20 | 11 | 56
Baseline lesions counts [Mean (Full Range); unit: lesions]
  Inflammatory lesions | 29.9 [20 to 74] | 29.0 [20 to 74] | 31.9 [20 to 72] | 28.6 [20 to 63] | 30.5 [20 to 75] | 30.0 [20 to 75]
  Non-inflammatory lesions | 43.5 [21 to 99] | 44.5 [21 to 98] | 46.7 [21 to 91] | 47.2 [20 to 98] | 43.9 [20 to 99] | 45.2 [20 to 99]

OUTCOME MEASURES:

1. Primary Outcome: Investigator's Global Assessment (IGA) "Success" - Week 12
Description: Count and percentage of subjects achieving success in each treatment group at Week 12 using the dichotomized IGA with success defined as a score of "clear" or "almost clear" (IGA Score of 0 or 1) and a two or more grade improvement from Baseline using a five-point scale (0=clear to 4=severe).
Time Frame: Baseline and Week 12
Population: Per-Protocol Population, defined as a subset of the ITT population and included those subjects that met eligibility criteria, completed the end-of-study visit, and applied at least 80% of the expected treatment applications.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose Active, BID | Medium-dose Active, BID | High-dose Active, QD | High-dose Active, BID | Vehicle, QD or BID
Number analyzed (Participants) | 57 | 64 | 52 | 55 | 59
Participants | 5 | 3 | 2 | 6 | 2

2. Primary Outcome: Inflammatory and Non-Inflammatory Lesion Counts - Week 12
Description: Absolute change from Baseline in inflammatory and non-inflammatory lesion counts in each treatment group at Week 12.
Time Frame: Baseline and Week 12
Population: Per protocol population.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Low-dose Active, BID | Medium-dose Active, BID | High-dose Active, QD | High-dose Active, BID | Vehicle, QD or BID
Number analyzed (Participants) | 55 | 62 | 52 | 55 | 57
lesions
  Inflammatory lesions | -8.3 (14.63) | -5.8 (11.99) | -10.1 (12.53) | -12.3 (14.43) | -9.1 (13.67)
  Non-inflammatory lesions | -8.7 (18.16) | -6.1 (29.22) | -8.4 (21.55) | -15.5 (20.48) | -6.7 (19.65)

3. Secondary Outcome: Inflammatory and Non-Inflammatory Lesion Counts - Week 8
Description: Absolute change from Baseline in inflammatory and non-inflammatory lesion counts in each treatment group at Week 8.
Time Frame: Baseline and Week 8
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Low-dose Active, BID | Medium-dose Active, BID | High-dose Active, QD | High-dose Active, BID | Vehicle, QD or BID
Number analyzed (Participants) | 54 | 62 | 52 | 53 | 56
lesions
  Inflammatory lesions | -11.9 (8.84) | -7.2 (12.03) | -7.2 (17.21) | -11.5 (11.19) | -11.3 (12.71)
  Non-inflammatory lesions | -7.0 (13.76) | -6.7 (16.33) | -3.2 (37.01) | -13.6 (17.99) | -8.3 (17.12)

4. Secondary Outcome: Percent Change in Lesion Counts - Weeks 8 and 12
Description: Percent change from Baseline in lesion counts (inflammatory and noninflammatory) in each treatment group at Weeks 8 and 12.
Time Frame: Week 8 and Week 12
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Low-dose Active, BID | Medium-dose Active, BID | High-dose Active, QD | High-dose Active, BID | Vehicle, QD or BID
Number analyzed (Participants) | 54 | 62 | 52 | 53 | 56
percentage of change
  Inflammatory lesions (Week 8) | -40.6 (28.20) | -26.6 (37.35) | -27.5 (41.44) | -41.1 (36.54) | -36.0 (35.01)
  Inflammatory lesions (Week 12) | -26.8 (50.78) | -21.3 (45.33) | -32.5 (35.51) | -41.8 (52.25) | -28.4 (41.88)
  Non-inflammatory lesions (Week 8) | -18.3 (34.50) | -19.5 (36.49) | -10.5 (57.13) | -33.5 (39.26) | -24.3 (43.23)
  Non-inflammatory lesions (Week 12) | -24.3 (38.69) | -16.9 (55.66) | -19.5 (40.75) | -34.1 (46.95) | -19.5 (47.43)

5. Secondary Outcome: IGA "Success" - Week 8
Description: Count and percentage of subjects achieving success per the IGA in each treatment group at Week 8 ("success" as defined in the primary endpoints section).
Time Frame: Baseline and Week 8
Population: Per protocol population.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose Active, BID | Medium-dose Active, BID | High-dose Active, QD | High-dose Active, BID | Vehicle, QD or BID
Number analyzed (Participants) | 54 | 62 | 52 | 53 | 56
Participants | 1 | 3 | 1 | 4 | 2

6. Secondary Outcome: IGA "Clear" or "Almost Clear" - Weeks 4, 8 and 12
Description: Count and percentage of subjects who are "clear" or "almost clear" (IGA Grade 0 or 1) in each treatment group at Weeks 4, 8 and 12.
Time Frame: Weeks 4, 8, and 12
Population: Per protocol population.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose Active, BID | Medium-dose Active, BID | High-dose Active, QD | High-dose Active, BID | Vehicle, QD or BID
Number analyzed (Participants) | 57 | 64 | 52 | 55 | 59
Participants
  Week 4: number analyzed (Participants) | 55 | 62 | 52 | 55 | 57
  Week 4 | 3 | 1 | 5 | 7 | 2
  Week 8: number analyzed (Participants) | 54 | 62 | 52 | 53 | 56
  Week 8 | 3 | 4 | 2 | 6 | 4
  Week 12 | 6 | 4 | 3 | 9 | 4

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from screening visit, Baseline (Day 1) and up to Week 12/early termination.
Arm/Group | Low-dose Active, BID | Medium-dose Active, BID | High-dose Active, QD | High-dose Active, BID | Vehicle, QD or BID
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/76 | 0/70 | 0/70 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/76 | 0/70 | 0/70 | 0/75
Other Adverse Events (participants affected / at risk) | 12/72 | 18/76 | 9/70 | 5/70 | 5/75
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose Active, BID (N=72) | Medium-dose Active, BID (N=76) | High-dose Active, QD (N=70) | High-dose Active, BID (N=70) | Vehicle, QD or BID (N=75)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 8 (8) | 2 (2) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has first right to publish pooled study data. In the event that such manuscript has not been submitted for publication within 18 months from study completion/termination at all participating sites, the PI shall have the right to single center publications provided they submit any data for presentation, oral or written, to the Sponsor for review 60 days prior to public disclosure. The PI may not disclose previously undisclosed confidential information other than study results.